CLINICAL TRIAL: NCT06219837
Title: Subarachnoid Block Versus Ultrasound Guided Transversalis Fascia Plane Block for Postoperative Analgesia of Inguinal Hernia Repair in Adults: A Randomized, Double Blinded, Controlled Trial
Brief Title: Subarachnoid Block Versus Ultrasound Guided Transversalis Fascia Plane Block for Postoperative Analgesia of Inguinal Hernia Repair in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rabab, lecture of anathesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: (TFP) block
Record Dates: First submitted 2023-06-06; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Analgesia of Inguinal Hernia Repair in Adults

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine group (Active Comparator): the patient in this arm will receive 20 ml of 0.25% bupivacaine injection by ultrasound guided transversalis fascia block for inguinal herniorraphy
  Interventions: Drug: bupivacaine injection by ultrasound guided transversalis fascia plane block
- 20 ml of 0.9% normal saline solution (Placebo Comparator): he patient in this arm will receive 20 ml of 0.9% normal saline solution by ultrasound guided transversalis fascia block for inguinal herniorraphy
  Interventions: Drug: bupivacaine injection by ultrasound guided transversalis fascia plane block

INTERVENTIONS:
Drug: bupivacaine injection by ultrasound guided transversalis fascia plane block — With patients in a sitting position and after appropriate skin asepsis, a 25-G pencil-point spinal needle (Pencil Point Spinal Needle Set, Egemen International Ltd., Izmir, Turkey) will be inserted through the L3 to L4 or L4 to L5 intervertebral space and 15 mg of 0.5% hyperbaric bupivacaine (AstraZeneca Pharmaceuticals, Cambridge, United Kingdom) will be injected. Subsequently, the patients will be positioned supine.
  Other Names: 20 ml of 0.9% normal saline solution

SUMMARY:
The aim of our study is to investigate the effect of the ultrasound guided transversalis fascia plane block on the postoperative opioid consumption as a part of multimodal analgesia in patients undergoing inguinal herniorrhaphy under spinal anesthesia.

DETAILED DESCRIPTION:
The aim of our study is to investigate the efficacy of the ultrasound-guided transversalis fascia plane block as a postoperative analgesia as a part of multimodal analgesia in patients undergoing inguinal herniorrhaphy under spinal anesthesia.

The ultrasound (US)-guided transversalis fascia plane (TFP) block was first described by Hebbard in 2009. A local anesthetic (LA) injected between the transversus abdominis muscle, and its deep investing fascia will block the anterior and the lateral branches of the T12 and L1 nerves (4). The efficacy of this block has been demonstrated in iliac crest bone graft harvesting, caesarean section and inguinal herniorrhaphy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing inguinal herniorrhaphy.
* Patients 18-60 years.
* ASA I and II.
* Both sexes.
* Having no contraindication for spinal anesthesia or TFP block.

Exclusion Criteria:

* Refusal of regional anesthesia.
* Infection in the back or at the site of injection for TFP block.
* INR > 1.5.
* Platelet count < 80000 per microliter of blood.
* Patients known to be allergic to amide local anesthetics.
* BMI greater than 35 kgm_2.
* Opioid addiction.
* Have communication problems that may hinder the assessement of pain postoperative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The total amount of postoperative morphine consumption during the first 24hrs postoperative. | First 24 hours postoperative
  The patients will be evaluated regarding the first demand to rescue analgesia postoperatively. The pain will be assessed by the VAS score. It will be performed in the immediate post-operative period every 15 min for the first 60 min, 2 h, 4 h, 8h, 12h, 18 and 24 h. Breakthrough pain will be defined as VAS >4 at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Zayed, Assistant professor, Study Director — Cairo University; Belal Khater, Master, Principal Investigator — Cairo University; Mohamed Mohamed, MD, Study Director — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Giza Governorate, Egypt